CLINICAL TRIAL: NCT05442528
Title: Six-month lead-in Study to Collect Prospective Efficacy and Safety Data of Current Replacement Therapy in Adult Hemophilia B Patients -- An Observational Survey Analysis Study
Brief Title: Lead-in Study of VGB-R04 Gene Therapy for Hemophilia B-- An Observational Survey Analysis Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: VGB-R04-LI
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: FIX replacement therapy.: Subject's previous treatment plan will be followed

SUMMARY:
This is a prospective, open, multicenter, observational lead-in study，to collect prospective efficacy and safety data of current replacement therapy in adult hemophilia B patients.

DETAILED DESCRIPTION:
Hemophilia B is a genetic bleeding disorder caused by pathogenic variants (eg, mutations, deletion) in the FIX gene. HB patients have frequent and potentially life-threatening bleeding and often develop progressive physical disability and pain from chronic haemarthropathy. Current replacement therapy needs regular treatment in the life-long time, bringing heavy economic and social burdens.VGB-R04 is a novel AAV vector carrying a high specific activity factor IX variant.

This is a prospective, open, multicenter, observational lead-in study. To evaluate the efficacy and safety of current treatment regiments in patients with moderate to severe HB (FIX:C activity ≤2%). The efficacy and safety data collected in this study may be used as baseline data for subsequent related clinical trials of VGB-R04. All subjects in this study will provide informed consent and then undergo screening assessments up to 4 weeks. All subjects will undergo 26 weeks of efficacy and safety observation .Eligible subjects will be invited to a key clinical study（phase 2 study）of VGB-R04,and then encouraged to enroll in an Long-term follow-up study to evaluate the long-term safety of VGB-R04 for a total of five years.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years and ≤65years of age;
2. Confirmed diagnosis of hemophilia B (baseline FIX activity ≤ 2% of normal);
3. At least 50 days exposure history to FIX;
4. Currently receiving FIX Prophylaxis therapy or on-demand treatment to prevent bleeding;
5. Have acceptable laboratory values:

   1. Hemoglobin ≥110 g/L;
   2. Platelets ≥100×109 /L;
   3. AST, ALT, alkaline phosphatase ≤2×upper limit of normal (ULN) at the testing laboratory;
   4. Bilirubin ≤3× ULN ;
   5. Creatinine ≤1.5× ULN.
6. No measurable factor IX inhibitor as assessed by the central laboratory and have no prior history of inhibitors to factor IX protein;

Exclusion Criteria:

1. Have significant underlying liver disease within the past 6 months prior to or at Screening, including but not limited to:

   1. Preexisting diagnosis of portal hypertension;
   2. Splenomegaly;
   3. Encephalopathy;
   4. Reduction of serum albumin;
   5. Evidence of significant liver fibrosis;
2. Have anti-VGB-R04 neutralizing antibody titers ≥1:5;
3. Evidence of severe infection disease, i.e., human immunodeficiency virus (HIV) infection, syphilis, tuberculosis, etc.;
4. Novel coronavirus infection occurred in the 6 weeks prior to entry into the group
5. Evidence of active hepatitis B virus infection (HBsAg positive) or hepatitis C virus infection (HCV-RNA positive);
6. Evidence of malignant tumours or those with a previous history of malignant tumours;
7. Have a history of chronic infection or other chronic diseases that the Investigator considers to constitute an unacceptable risk;
8. Any immunodeficiency;
9. planned surgery may be required within one year;
10. Past thromboembolic events (arterial or venous thromboembolic events);
11. Hypertensive patients with poor blood pressure control (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90mmHg after antihypertensive drug treatment);

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemophilia B (baseline FIX activity ≤ 2% of normal)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate changes from baseline | Baseline up to Week 26
  The number of bleeding episodes per participant will be recorded, and the annualized number of bleeding episodes.

SECONDARY OUTCOMES:
Annualized FIX consumption changes from baseline | Baseline up to Week 26
  The use of on-demand FIX replacement therapy will be recorded by dose (IU/kg) administered, and the annualized use of FIX replacement therapy will be calculated.
Total number of annualized bleeding | Baseline up to Week 26
  Total number of annualized bleeding including spontaneous or traumatic bleeding.
FIX:C activity level. | Baseline up to Week 26
  FIX:C activity level and its change from baseline .
Number of target joints | Baseline up to Week 26
  The criterion of the target joint is a minimum of three bleeds into a single joint within a consecutive three-month period.
The incidence of adverse Events of special interest | Baseline up to Week 26
  Adverse Events of special interest (serious or non-serious) are a category of events of scientific and medical concern that are particularly relevant to the sponsor's drug or research program. Adverse Events of special interest include liver dysfunction, inhibitors, thromboembolic events, and allergic reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGB-R04 is fully approved.
Time Frame: IPD will be shared with other researchers when VGB-R04 is fully approved.
Access Criteria: IPD will be shared with other researchers when VGB-R04 is fully approved.